CLINICAL TRIAL: NCT03495596
Title: Determination of Factors Leading to Failure of Videolaryngoscopy
Brief Title: Predictors of Difficult Videolaryngoscopy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sevilay Kivrakoglu, HacettepeU, Hacettepe University
Other Study IDs: Videolaryngoscopy
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Videolaryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Videolaryngoscopy patients: The patients who were attempted to be intubated with videolaryngoscopy
  Interventions: Device: Videolaryngoscopy

INTERVENTIONS:
Device: Videolaryngoscopy — Videolaryngoscopy device type

SUMMARY:
The primary goal of this study was to identify parameters affecting the failure of videolaryngoscopy in clinical practice; secondly, the incidence of videolaryngoscopy use and the most frequently used patient groups.

DETAILED DESCRIPTION:
Videolaryngoscopy is widely used in the management of patients with presumed difficult airway. It offers an improved laryngeal view compared with direct laryngoscopy and increases the likelihood of successful intubation in patients for whom direct laryngoscopy is anticipated to be difficult. It is among the most frequently preferred difficult airway devices due to its ease of use, portability and direct laryngoscopy resemblance. The use of videolaryngoscopy has been shown to improve intubation success in many cases associated with difficult intubation, such as morbid obesity, pregnancy, limitation of cervical motility, and poor mouth opening.

ELIGIBILITY:
Inclusion Criteria:

* All patients who used videolaryngoscopy for intubation

Exclusion Criteria:

-

Ages: 1 Day to 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will undergo surgery under general anesthesia will be followed in Hacettepe University Hospital's operating room. All patients aged 0-95 years who used videolaryngoscopy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1159 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Intubation success | 15 minutes
  The success of intubation attempt with videolaryngoscopy (yes/no)

SECONDARY OUTCOMES:
The reason of videolaryngoscopy | 15 minutes
  Why videolaryngoscopy is preferred instead of standard direct laryngoscopy
The type of videolaryngoscopy blade | 15 minutes
  acute angled/macintosh/miller blade
The rescue technique | 30 minutes
  The rescue technique used for patients who could not be intubated with videolaryngoscopy
Factors affecting success of videolaryngoscopy | 30 minutes
  Mallampati score, thyromental distance, neck movements, upper lip bite test, mouth opening

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Ankay Yilbas, MD, Study Director — Turkish Society of Anesthesiology and Reanimation; Sevilay Kivrakoglu, MD, Principal Investigator — Turkish Society of Anesthesiology and Reanimation
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Aziz MF, Bayman EO, Van Tienderen MM, Todd MM; StAGE Investigator Group; Brambrink AM. Predictors of difficult videolaryngoscopy with GlideScope(R) or C-MAC(R) with D-blade: secondary analysis from a large comparative videolaryngoscopy trial. Br J Anaesth. 2016 Jul;117(1):118-23. doi: 10.1093/bja/aew128. PMID 27317711
- [Background] el-Ganzouri AR, McCarthy RJ, Tuman KJ, Tanck EN, Ivankovich AD. Preoperative airway assessment: predictive value of a multivariate risk index. Anesth Analg. 1996 Jun;82(6):1197-204. doi: 10.1097/00000539-199606000-00017. PMID 8638791
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Toshniwal G, McKelvey GM, Wang H. STOP-Bang and prediction of difficult airway in obese patients. J Clin Anesth. 2014 Aug;26(5):360-7. doi: 10.1016/j.jclinane.2014.01.010. Epub 2014 Jul 28. PMID 25081584
- [Background] Nakao K, Komasawa N, Kusaka Y, Minami T. Rapid-Sequence Intubation in the Left-Lateral Tilt Position in a Pregnant Woman with Premature Placental Abruption Utilizing a Videolaryngoscope. AJP Rep. 2015 Apr;5(1):e30-2. doi: 10.1055/s-0034-1544109. Epub 2015 Feb 25. PMID 26199794
- [Background] Kleine-Brueggeney M, Greif R, Schoettker P, Savoldelli GL, Nabecker S, Theiler LG. Evaluation of six videolaryngoscopes in 720 patients with a simulated difficult airway: a multicentre randomized controlled trial. Br J Anaesth. 2016 May;116(5):670-9. doi: 10.1093/bja/aew058. PMID 27106971
- [Background] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773
- [Background] Wilson ME, Spiegelhalter D, Robertson JA, Lesser P. Predicting difficult intubation. Br J Anaesth. 1988 Aug;61(2):211-6. doi: 10.1093/bja/61.2.211. PMID 3415893
- [Background] Nath G, Sekar M. Predicting difficult intubation--a comprehensive scoring system. Anaesth Intensive Care. 1997 Oct;25(5):482-6. doi: 10.1177/0310057X9702500505. PMID 9352759
- [Background] Benumof JL. Management of the difficult adult airway. With special emphasis on awake tracheal intubation. Anesthesiology. 1991 Dec;75(6):1087-110. doi: 10.1097/00000542-199112000-00021. PMID 1824555
- [Background] Williamson JA, Webb RK, Szekely S, Gillies ER, Dreosti AV. The Australian Incident Monitoring Study. Difficult intubation: an analysis of 2000 incident reports. Anaesth Intensive Care. 1993 Oct;21(5):602-7. doi: 10.1177/0310057X9302100518. PMID 8273882
- [Background] Nichol HC, Zuck D. Difficult laryngoscopy--the "anterior" larynx and the atlanto-occipital gap. Br J Anaesth. 1983 Feb;55(2):141-4. doi: 10.1093/bja/55.2.141. PMID 6830676
- [Background] Oates JD, Macleod AD, Oates PD, Pearsall FJ, Howie JC, Murray GD. Comparison of two methods for predicting difficult intubation. Br J Anaesth. 1991 Mar;66(3):305-9. doi: 10.1093/bja/66.3.305. PMID 2015145
- [Background] Charters P, Perera S, Horton WA. Visibility of pharyngeal structures as a predictor of difficult intubation. Anaesthesia. 1987 Oct;42(10):1115. doi: 10.1111/j.1365-2044.1987.tb05182.x. No abstract available. PMID 3688398
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827